## 12/21/2017

Study: Excess Opioid Disposal Following Orthopedic Foot and Ankle Surgery

NCT03285061

**Statistical Analysis Plan** 

## 12/21/2017

## Study: Excess Opioid Disposal Following Orthopedic Foot and Ankle Surgery NCT03285061

## **Statistical Analysis Plan**

We aim to enroll at least 35 patients in each group assuming a follow-up rate to study completion of approximately 60%. Treatment groups are to be compared using a Chi-Square Test of Independence. P-values less than 0.05 are to be considered statistically significant. All statistical analyses are to be conducted using R and Microsoft Excel (R Project, Microsoft Corporation).